CLINICAL TRIAL: NCT03485027
Title: A Phase II Clinical Trial of Prior Regimen Rechallenge in Third or Later-line Chemotherapy for Patients With Metastatic Colorectal Cancer
Brief Title: Rechallenge of Prior Regimen in Third or Later-line Chemotherapy in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Weijian Guo, Vice director of Dep.Medical Oncology, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-RC
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Colorectal Cancer; Chemotherapy Effect
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: investigator chose the optimal reintroduction regimen for chemotherapy according to criteria
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The rechallenge regimens (Experimental): XELOX ± BEV, repeating every 3 weeks.
  FOLFOX ± BEV, repeating every 2 week
  FOLFOX ± Cetuximab, repeating every 2 week
  FOLFIRI ± BEV, repeating every 2 weeks.
  FOLFIRI ± Cetuximab, repeating every 2 weeks.
  IRI ± BEV, repeating every 2 weeks.
  IRI ± Cetuximab, repeating every 2 weeks.
  Raltitrexed ± BEV, repeating every 3 weeks.
  Raltitrexed ± Cetuximab, repeating every 2 weeks.
  Interventions: Drug: the rechallenge regimen

INTERVENTIONS:
Drug: the rechallenge regimen — XELOX regimen: Oxaliplatin 130mg/m2, intravenous, on day 1; Capecitabine 1000mg/m2, oral, twice daily, continuously for 14 days; ±bevacizumab 7.5mg/kg, intravenous, on day 1; repeating every 3 weeks. FOLFOX regimen: Oxaliplatin 85mg/m2 on day 1; Calcium folinate 400mg/m2 on day 1; 5-FU 400mg/m2 on day 1; 5-FU 2.4g/m2, continuous intravenous infusion for 46 hours, ± Bevacizumab 5mg/kg or ± Cetuximab 500mg/m2, repeating every 2 weeks. FOLFIRI regimen: Irinotecan 180mg/m2 on day 1; Calcium folinate 400mg/m2 on day 1; 5-FU 400mg/m2 on day 1; 5-FU 2.4g/m2, continuous intravenous infusion for 46 hours; ± Bevacizumab 5mg/kg or ± Cetuximab 500mg/m2, repeating every 2 weeks. Irinotecan monotherapy regimen: Irinotecan 180mg/m2 on day 1, ± Bevacizumab 5mg/kg or ± Cetuximab 500mg/m2, repeating every 2 weeks. Raltitrexed contained regimen: Raltitrexed 3mg/m2 on day 1; ± Bevacizumab 7.5mg/kg, repeating every 3 weeks; Raltitrexed 2mg/m2 on day 1; ± Cetuximab 500mg/m2, repeating every 2 weeks.
  Other Names: reintroduction of the former regimens in the third or later line treatment even after the same treatment had shown drug-resistance in the former setting

SUMMARY:
This is a single-arm, open-label, single-center prospective phase II study to evaluate the efficacy and safety of rechallenge chemotherapy in the third or later-line treatment in patients with advanced colorectal cancer. The primary end point is progression free survival (PFS). A total of 42 patients who failed with oxaliplatin, irinotecan and fluorouracil in previous treatment and could not receive the target therapy presently are planned for recruitment. For patients with metastatic colorectal cancer who met admission criteria, oxaliplatin- or irinotecan-based chemo regimen could be used and evaluation was repeated every 6 weeks. The treatment continues until the disease progression or the untolerable adverse reaction.

DETAILED DESCRIPTION:
The treatment for reintroduction was oxaliplatin- or irinotecan-based chemo-regimen.

Optional chemotherapy regimen included XELOX,FOLFOX,FOLFIRI,Irinotecan single-agent

ELIGIBILITY:
Inclusion Criteria

1. Patients age between 18 and 80 years
2. Histologically confirmed metastatic colorectal cancer (mCRC)
3. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
4. Treatment failure to at least two lines of chemotherapy (regimens should include oxaliplatin, fluorouracil and irinotecan); progression free survival (PFS) of prior oxaliplatin or irinotecan-based chemotherapy should be at least four months without any unrecoverable toxicity. Prior target therapy was acceptable
5. For those who received other anti-tumor treatment, the toxicity should have been restored, with the time interval from last dose of cytotoxic drugs, radiation or surgery (the wound should be healed completely) ≥3 weeks
6. Life expectancy≥12 weeks
7. At least one measurable lesion as defined by RECIST 1.1
8. Acceptable hematologic, hepatic, and renal function within 7 days from screening: the blood ANC count≥1.5*10^9/L; hemoglobin≥9.0 g/dl, the blood platelet count≥80 x 10^9/L, total bilirubin<1.5*upper limits of normal(ULN), ALT and AST<2.5*ULN(< 5 *ULN for patients with live metastasis), endogenous creatinine clearance rate>50ml/min
9. Targeted drugs are currently not suitable or affordable

Exclusion Criteria

1. Receiving other systemic anti-cancer treatment within 3 weeks
2. Prior radiation therapy of target measurable lesion
3. Presence of Grade III or IV chemo-related toxicity in previous treatment without recovery to Grade II or less
4. With other malignant tumor in 5 years; except for cured cervical carcinoma in situ or basal cell carcinoma
5. Symptomatic intracranial or meningeal metastasis
6. History of uncontrolled seizures, central nervous system dysfunction or mental disorder
7. Uncontrolled pleural or peritoneal effusion
8. Severe life-threatening concomitant disease that might impair the safety of patients or affect the completion of treatment, according to the researcher's judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
PFS | from the time signing of informed consent form(ICF) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  progression free survival

SECONDARY OUTCOMES:
OS | from the time signing of ICF until the date of death from any cause, assessed up to 48 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided